CLINICAL TRIAL: NCT02017535
Title: A Personalized Approach to Achieving a Sustained Response to Treatment for Adolescent Depression
Brief Title: An Adaptive Treatment Strategy for Adolescent Depression-Continuation
Acronym: PTAD GIA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1206M15365
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Adolescent Depression
MeSH Terms: interventions — Fluoxetine; Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 6 IPT-A Sessions (Active Comparator): Participants in this group will receive interpersonal psychotherapy for adolescents (IPT-A) only.
  During the Continuation IPT-A sessions, the therapist will continue to emphasize the interpersonal strategies that were learned and practiced during the acute phase, and address any current interpersonal problems before they result in a recurrence of depressive symptoms. Adolescents who have responded to acute phase treatment (CGI-I = much improved or very much improved) will attend 4 biweekly IPT-A sessions followed by 2 monthly sessions.
  Interventions: Behavioral: Interpersonal Psychotherapy
- 6 IPT-A Sessions + Continue Current Dose of Fluoxetine (Active Comparator): Participants in this group will receive interpersonal psychotherapy for adolescents (IPT-A) and fluoxetine treatment.
  Adolescents who have responded to acute phase treatment (CGI-I = much improved or very much improved) will attend 4 biweekly IPT-A sessions followed by 2 monthly sessions and will continue their acute phase fluoxetine dosing regimen and will meet with the psychiatrist on a monthly basis.
  Interventions: Drug: Fluoxetine; Behavioral: Interpersonal Psychotherapy
- 10 IPT-A Sessions + Begin Fluoxetine (Experimental): Participants in this group will receive interpersonal psychotherapy for adolescents (IPT-A) and fluoxetine treatment.
  Adolescents who received only IPT-A during acute phase and who showed a partial response (CGI-I = minimally improved) will attend 8 weekly IPT-A sessions followed by 2 monthly sessions and will begin treatment with fluoxetine during the continuation phase.The dosage schedule will be 10mg per day for the first week and 20mg per day for the following 5 weeks. If no treatment response is observed by the 6th week, the dosage can be increased to 40mg per day. Pharmacotherapy sessions will be scheduled weekly for the first 4 weeks and biweekly thereafter. Pharmacotherapy sessions will include assessment of vital signs, adverse effects, safety, and symptomatic response.
  Interventions: Drug: Fluoxetine; Behavioral: Interpersonal Psychotherapy
- 10 IPT-A Sessions + Increase Dose of Fluoxetine (Experimental): Participants in this group will receive interpersonal psychotherapy for adolescents (IPT-A) and fluoxetine treatment.
  Adolescents who received IPT-A and fluoxetine during the acute phase and were partial responders (CGI-I = minimally improved) will attend 8 weekly IPT-A sessions followed by 2 monthly sessions and will have their fluoxetine dose increased to 60mg. Partial responders will meet with the psychiatrist biweekly for the first 2 months and monthly for the second 2 months.
  Interventions: Drug: Fluoxetine; Behavioral: Interpersonal Psychotherapy

INTERVENTIONS:
Drug: Fluoxetine — Prozac (fluoxetine capsules, USP) is a selective serotonin reuptake inhibitor for oral administration.
  Other Names: Prozac
  Arms: 10 IPT-A Sessions + Begin Fluoxetine; 10 IPT-A Sessions + Increase Dose of Fluoxetine; 6 IPT-A Sessions + Continue Current Dose of Fluoxetine
Behavioral: Interpersonal Psychotherapy — Type of talk therapy that focuses on an adolescents relationship and communication skills in the context of of their depression.
  Other Names: IPT

SUMMARY:
Aim 1: Assess the feasibility and acceptability of the personalized continuation treatment strategy.

Aim 2: Estimate variances of primary and secondary outcomes with the continuation treatment.

Aim 3: Conduct exploratory hypothesis-generating analyses to inform further development of the personalized continuation treatment strategy to be tested in a subsequent R01 proposal.

DETAILED DESCRIPTION:
Male and female adolescents (ages 12-18) will be eligible for the study if they completed acute phase treatment and showed at least a partial response to treatment (CGI-I of minimally improved or better (CGI-I < 3)). Adolescents will enter continuation treatment having either received 12 sessions of IPT-A, 16 sessions of IPT-A, or 12 sessions of IPT-A plus fluoxetine.This is a continuation of the study "An Adaptive Treatment Strategy for Adolescent Depression (PTAD)" NCT01802437

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and parents must be English-speaking
* Completed acute phase treatment (NCT01802437) and showed at least a partial response to treatment (CGI-I of minimally improved or better (CGI-I < 3)).

Exclusion Criteria:

- Did not completed acute phase treatment (NCT01802437) or did not show at least a partial response to treatment (CGI-I of minimally improved or better (CGI-I < 3)) to acute phase treatment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Gunlicks-Stoessel, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Department of Psychiatry, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Gunlicks-Stoessel M, Mufson L, Bernstein G, Westervelt A, Reigstad K, Klimes-Dougan B, Cullen K, Murray A, Vock D. Critical Decision Points for Augmenting Interpersonal Psychotherapy for Depressed Adolescents: A Pilot Sequential Multiple Assignment Randomized Trial. J Am Acad Child Adolesc Psychiatry. 2019 Jan;58(1):80-91. doi: 10.1016/j.jaac.2018.06.032. Epub 2018 Oct 27. PMID 30577943

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 IPT-A Sessions: IPT Only
  Interpersonal Psychotherapy (IPT): Type of talk therapy that focuses on an adolescents relationship and communication skills in the context of of their depression.
- 6 IPT-A Sessions + Continue Current Dose of Fluoxetine: IPT with continued current fluoxetine dosage
  Interpersonal Psychotherapy (IPT): Type of talk therapy that focuses on an adolescents relationship and communication skills in the context of of their depression.
  Fluoxetine: Adolescents who receive pharmacotherapy will be prescribed fluoxetine for 12 weeks. The dosage schedule will be 10 mg per day for the first week and 20 mg per day for the following 5 weeks. If no treatment response is observed by week 6, the dosage can be increased to 40 mg per day. Pharmacotherapy sessions will be scheduled weekly for the first 4 weeks and every other week thereafter.
- 10 IPT-A Sessions + Begin Fluoxetine: IPT with new fluoxetine use
  Interpersonal Psychotherapy (IPT): Type of talk therapy that focuses on an adolescents relationship and communication skills in the context of of their depression.
  Fluoxetine: Adolescents who receive pharmacotherapy will be prescribed fluoxetine for 12 weeks. The dosage schedule will be 10 mg per day for the first week and 20 mg per day for the following 5 weeks. If no treatment response is observed by week 6, the dosage can be increased to 40 mg per day. Pharmacotherapy sessions will be scheduled weekly for the first 4 weeks and every other week thereafter.
- 10 IPT-A Sessions + Increase Dose of Fluoxetine: IPT with increased dose of fluoxetine
  Interpersonal Psychotherapy (IPT): Type of talk therapy that focuses on an adolescents relationship and communication skills in the context of of their depression.
  Fluoxetine: Adolescents who receive pharmacotherapy will be prescribed fluoxetine for 12 weeks. The dosage schedule will be 10 mg per day for the first week and 20 mg per day for the following 5 weeks. If no treatment response is observed by week 6, the dosage can be increased to 40 mg per day. Pharmacotherapy sessions will be scheduled weekly for the first 4 weeks and every other week thereafter.
Period: Overall Study
Arm/Group | 6 IPT-A Sessions | 6 IPT-A Sessions + Continue Current Dose of Fluoxetine | 10 IPT-A Sessions + Begin Fluoxetine | 10 IPT-A Sessions + Increase Dose of Fluoxetine
Started | 9 | 3 | 2 | 1
Completed | 8 | 3 | 2 | 1
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 IPT-A Sessions | 6 IPT-A Sessions + Continue Current Dose of Fluoxetine | 10 IPT-A Sessions + Begin Fluoxetine | 10 IPT-A Sessions + Increase Dose of Fluoxetine | Total
Number analyzed (Participants) | 8 | 3 | 2 | 1 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 3 | 2 | 1 | 14
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.25 (1.91) | 15 (1.73) | 13 (1.41) | 16 (NA) — Single participant, SD cannot be calculated. | 14.93 (1.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 1 | 1 | 11
  Male | 1 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 2 | 2 | 0 | 11
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 2 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Children's Depression Rating Scale-Revised (CDRS-R)
Description: The CDRS-R is a clinician-administered semi-structured interview designed to assess present episode and lifetime history of psychiatric diagnoses based on DSM-IV criteria. This survey contains 17 items; 3 items are rated on a scale from 0 to 5, 5 items are rated on a scale from 0 to 6, and the remaining 9 items are rated on a scale from 0 to 7. Total score is a raw sum of the 17 item scores and ranges from 0 to 108. Higher scores indicate greater depression severity.
Time Frame: 16 weeks, 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 6 IPT-A Sessions | 6 IPT-A Sessions + Continue Current Dose of Fluoxetine | 10 IPT-A Sessions + Begin Fluoxetine | 10 IPT-A Sessions + Increase Dose of Fluoxetine
Number analyzed (Participants) | 8 | 3 | 2 | 1
score on a scale
  16 Weeks | 32.38 (7.31) | 26.67 (7.23) | 51 (4.24) | 45 (NA) — Only one participant in this group, standard deviation can not be calculated.
  32 Weeks | 29 (7.07) | 33.33 (5.51) | 29 (9.9) | 51 (NA) — Only one participant in this group, standard deviation can not be calculated.

2. Primary Outcome: Children's Global Assessment Scale (CGAS)
Description: The CGAS is a numeric scale used by mental health clinicians to rate the general functioning of youths under the age of 18. Scores range from 1 to 100, with higher scores indicating better functioning.
Time Frame: 16 weeks, 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 6 IPT-A Sessions | 6 IPT-A Sessions + Continue Current Dose of Fluoxetine | 10 IPT-A Sessions + Begin Fluoxetine | 10 IPT-A Sessions + Increase Dose of Fluoxetine
Number analyzed (Participants) | 8 | 3 | 2 | 1
score on a scale
  16 weeks | 65 (4) | 77 (8) | 53 (4) | 55 (NA) — Only one participant in this group, standard deviation can not be calculated.
  32 weeks | 72 (10) | 71 (10) | 72 (5) | 49 (NA) — Only one participant in this group, standard deviation can not be calculated.

3. Primary Outcome: Beck Depression Inventory-II (BDI-II)
Description: BDI-II is a 21-item self-report multiple-choice inventory that assesses the severity of depressive symptoms reflective of DSM-IV diagnostic criteria over the prior week. Items are rated on a 4-point scale ranging from 0 to 3. Total scores are a sum of the 21 item scores ranging from 0 to 63. Higher scores indicate more severe depression symptoms.
Time Frame: 16 weeks, 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 6 IPT-A Sessions | 6 IPT-A Sessions + Continue Current Dose of Fluoxetine | 10 IPT-A Sessions + Begin Fluoxetine | 10 IPT-A Sessions + Increase Dose of Fluoxetine
Number analyzed (Participants) | 8 | 3 | 2 | 1
score on a scale
  16 weeks | 7.63 (4.27) | 11.33 (12.66) | 10 (14.14) | NA (NA) — Only one participant in this group; data point is missing.
  32 weeks | 5.86 (3.67) | 9 (10.82) | 1.5 (2.12) | 41 (NA) — Only one participant in this group; data point is missing.

4. Primary Outcome: Social Adjustment Scale - Self Report (SAS-SR)
Description: The SAS-SR is a 42-item self report measure of role performance in the past 2 weeks. Items are rated on a 5-point scale. Total scores are calculated by summing the 42 item scores and dividing by the total number of items answered. Total scores range from 1 to 5, with higher scores indicating greater impairment of functioning.
Time Frame: 16 weeks, 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 6 IPT-A Sessions | 6 IPT-A Sessions + Continue Current Dose of Fluoxetine | 10 IPT-A Sessions + Begin Fluoxetine | 10 IPT-A Sessions + Increase Dose of Fluoxetine
Number analyzed (Participants) | 8 | 3 | 2 | 1
score on a scale
  16 weeks | 2.03 (.49) | 2.07 (.22) | 2.75 (.67) | NA (NA) — Only one participant in this group; data point is missing.
  32 weeks | 2.17 (.55) | 1.62 (.46) | 2.18 (.17) | 3.09 (NA) — Only one participant in this group; data point is missing.

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | 6 IPT-A Sessions | 6 IPT-A Sessions + Continue Current Dose of Fluoxetine | 10 IPT-A Sessions + Begin Fluoxetine | 10 IPT-A Sessions + Increase Dose of Fluoxetine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT02017535/Prot_SAP_000.pdf